CLINICAL TRIAL: NCT04718480
Title: A Randomized, Double-blind, Placebo-controlled, Adaptive-design Study to Assess the Safety and Efficacy of Daily 200 mg Fluvoxamine as add-on Therapy to Standard of Care in Moderate Severity COVID-19 Patients
Brief Title: Fluvoxamine Administration in Moderate SARS-CoV-2 (COVID-19) Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SigmaDrugs Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SD-COVID19-01; 2020-002299-11 (EudraCT Number)
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: moderate COVID-19; fluvoxamine
MeSH Terms: conditions — COVID-19 | interventions — Fluvoxamine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, adaptive design add-on treatment study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo-controlled,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 2 x 100 mg placebo daily po. (with careful dose escalation and tapered dose reduction). Overall treatment period is 74 days.
  Interventions: Drug: Placebo
- Fluvoxamine (Experimental): 2 x 100 mg fluvoxamine daily po. (with careful dose escalation and tapered dose reduction). Overall treatment period is 74 days.
  Interventions: Drug: Fluvoxamine

INTERVENTIONS:
Drug: Placebo — po placebo tablets
  Arms: Placebo
Drug: Fluvoxamine — po fluvoxamine tablets
  Arms: Fluvoxamine

SUMMARY:
This is a randomized, double-blind, placebo-controlled, adaptive two-stage design, human phase 2 study, with add-on treatment arrangement of fluvoxamine or placebo on top of standard of care (base therapy: the actual proposed therapy of moderate SARS-CoV-2 infected patients according to "Hungarian Coronavirus Handbook", including antiviral and immunmodulant therapy and reconvalescent plasma therapy in serious cases as indicated by the investigator).

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-70 years of age at screening
* Hospitalized patients with confirmed SARS-CoV-2 by PCR or known contact of confirmed case with syndrome consistent with coronavirus disease (COVID-19) with PCR pending (positive PCR result should be available prior to randomisation).
* Moderate cases (each of the followings met): showing dyspnoea but not manifest respiratory distress, respiratory rate 22-29 / min; oxygen saturation at rest > 93%; with or without the need for oxygen supplementation; pneumonia on medical imaging with pulmonary infiltrates occupying ≤ 50% of the lung-fields
* Subjects who are able to communicate with the Investigator and research staff, who understand the study, are able to comply with all study procedures, and willing to provide written informed consent prior to the screening examinations.

Exclusion Criteria:

* Mild COVID-19 at randomisation (each of the followings met): no dyspnoea, respiratory rate < 22 / min, no need for oxygen supplementation, no pneumonia on medical imaging

  * Severe COVID-19 at randomisation: respiratory distress - respiratory rate ≥ 30/min, oxygen saturation at rest ≤ 93%, pulmonary infiltrates occupy > 50% of the lung-fields
  * Critical COVID-19 at randomisation: acute respiratory distress, requiring mechanical ventilation, radiomorphology of ARDS, shock, including septic shock, other organ dysfunction necessitating ICU admission
  * High-risk patient for progression of COVID-19, as defined by having a calculated pneumonia PORT-score of > 90
  * Concomitant or previous administration of any experimental, non-established COVID-19 therapy, either in off-label indication (of a registered medicinal product) or as a non-registered drug candidate in a clinical trial setting or compassionate use program (or equivalents thereof), EXCEPT therapies recommended by the "Magyar Koronavírus Kézikönyv" (Hungarian Coronavirus Manual), and as such, are considered as standard-of-care. Concomitant use of LMWHs can be considered as emerging standard-of-care, and therefore their application is not prohibited.
  * Standard of care treatment planned with chloroquine or hydroxychloroquine.
  * Any clinically significant abnormality identified during pre-study full physical examination, vital signs, laboratory tests and ECG which is deemed by the Investigator to be incompatible / inappropriate for study participation.
  * Known hepatitis B, C, or HIV infection.
  * A current or recent history of drug or substance abuse, including alcohol (> 14 units per week), within 3 months prior to screening (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or one shot [25 mL] of spirits)
  * Patients who regularly consume more than 4 cups daily of beverage containing caffeine
  * Current strong smoker as defined by smoking over 10 cigarettes a day, or its equivalent
  * Positive pregnancy test result for women with childbearing potential at screening
  * Women who are pregnant or nursing, or who are planning to get pregnant within 3 months after the last dose of study drug
  * A history of allergy, intolerance or sensitivity to fluvoxamine or any component of the study drug formulation
  * Closed-angle glaucoma
  * Patients who are assessed as at risk for suicidal intent during screening by psychiatric evaluation (including C-SSRS questionnaire). A score of 15 or higher on the PHQ-9 depression scale at screening.
  * Have undergone surgery or have donated blood within 12 weeks prior to the start of the study
  * A history of bleeding diathesis or other bleeding disorders
  * Participated in any clinical trial involving an investigational drug or investigational device within 1 month preceding study entry, or within 5 terminal half-life of the investigational drug of this previous study
  * A history of or present malignancy, with the exception of resected basal cell carcinoma or squamous cell carcinoma of the skin, or resected cervical intraepithelial neoplasia.

Prohibited concomitant medications:

* Co-administration of fluvoxamine with monoamine oxidase inhibitors (MAOI), including methylene blue (intravenous dye) and linezolid (an antibiotic which is a reversible non-selective MAOI)
* Co-administration of thioridazine, mesoridazine, pimozide, terfenadine, astemizole, or cisapride with fluvoxamine; each of these drugs alone produces prolongation of the QTc interval, which is associated with serious ventricular arrhythmias, such as torsade de pointes-type arrhythmias and sudden death
* Co-administration of tizanidine and fluvoxamine
* Co-administration of fluvoxamine with ramelteon
* Co-administration of fluvoxamine with chloroquine or hydroxychloroquine
* Co-administration of morphine, or other opioids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Time to clinical recovery after treatment | 74 days
  days from randomization (Day 1) to ANY THREE items of the following four:
  1. resolution from fever (oral or tympanic temperature ≤ 37.5 °C, axillary ≤ 37.0 °C for at least 48 hours without antipyretics)
  2. return of respiratory rate to normal (≤ 20 / min)
  3. normalization of SpO2 ( ≥95% on room air )
  4. cough remission (any reduction in cough-burden Visual Analogue Scale, compared to Day 1 baseline)

CONTACTS AND LOCATIONS:
Locations (4):
- Hungary (4):
  - Dél-pesti Centrumkórház, Budapest
  - Semmelweis Egyetem Pulmonológiai Klinika, Budapest
  - Országos Korányi Pulmonológiai Intézet, Budapest
  - Debreceni Egyetem Kenézy Gyula Kórház Infektológia, Debrecen

IPD SHARING:
Plan to Share IPD: No
Study results will be published at the end of the study.